CLINICAL TRIAL: NCT03089398
Title: Randomized Trial Of Hybrid Coronary Revascularization Versus Percutaneous Coronary Intervention
Brief Title: Hybrid Coronary Revascularization Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emilia Bagiella (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Emilia Bagiella, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 14-0250; 1U01HL125506-01A1 (NIH); 1U01HL125488-01A1 (NIH)
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: Hybrid Coronary Revascularization; Coronary Artery Bypass Grafting; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: This trial is a prospective, multi-center randomized comparative effectiveness trial of HCR compared to multi-vessel PCI with metallic DES in patients with multi-vessel CAD involving the LAD or LM territories.
Who Masked: Outcomes Assessor
Masking Description: The DCC Research Coordinator will be blinded to treatment assignment during follow-up telephone calls and will be blinded to aggregate outcomes data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Hybrid Coronary Revascularization Group (Active Comparator): HCR is defined, for the purposes of this trial, as a planned off-pump minimally invasive (sternal-sparing), isolated LIMA-LAD revascularization, combined with percutaneous revascularization of at least one non-LAD target.
  Interventions: Procedure: Hybrid Coronary Revascularization (isolated LIMA-LAD); Device: Hybrid Coronary Revascularization (PCI)
- Percutaneous Coronary Intervention (Active Comparator): PCI will be performed using standard techniques at the discretion of the operator. Only Food and Drug Administration (FDA) and Health Canada approved commercially available metallic drug-eluting stents may be used in this protocol.
  Interventions: Device: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Hybrid Coronary Revascularization (isolated LIMA-LAD) — sternal-sparing, off-pump, isolated LIMA-LAD revascularization
  Other Names: Left Internal Mammary Artery (LIMA) to LAD
  Arms: Hybrid Coronary Revascularization Group
Device: Hybrid Coronary Revascularization (PCI) — percutaneous revascularization of at least one non-LAD target
  Other Names: PCI with metallic DES of non-LAD vessel(s)
  Arms: Hybrid Coronary Revascularization Group
Device: Percutaneous Coronary Intervention — Multi-vessel PCI with metallic drug-eluting stents (DES) including the LAD and or LM. Only FDA approved commercially available metallic drug-eluting stents may be used in this protocol.
  Other Names: PCI
  Arms: Percutaneous Coronary Intervention

SUMMARY:
The purpose of the study is to learn which treatment option is better for patients who have multi-vessel coronary artery disease (blockages in more than one vessel supplying blood to the heart muscle). The treatment options this study will compare are: (1) Hybrid Coronary Revascularization [HCR] (a combination of surgery and catheter procedures to open up clogged heart arteries) and (2) Percutaneous Coronary Intervention [PCI] (catheter procedures alone to open up clogged heart arteries). There are no new or "experimental" procedures being tested in this study: both HCR and PCI are well-established procedures and are regularly performed in patients who have coronary artery disease. But, the FDA has not approved the drug-eluting stents used in PCI for all types of coronary artery disease. We have received an Investigational Device Exemption from the FDA to use the drug-eluting stents in this trial in the same way that they are used in clinical practice. The study being proposed here will use rigorous scientific methods and should result in a very high level of certainty about which procedure is best for patients with coronary artery disease.

DETAILED DESCRIPTION:
The increasing prevalence of coronary artery disease (CAD), advances in coronary artery bypass grafting (CABG), percutaneous coronary intervention (PCI), and concomitant medical therapy, and the costs of revascularization have resulted in rising interest regarding the appropriate indications and alternatives for coronary revascularization.

Hybrid coronary revascularization is the intended combination of CABG and PCI. The HCR strategy combines grafting of the left anterior descending artery (LAD) coronary artery using the left internal mammary artery (LIMA) and PCI of non-LAD coronary stenoses. Essentially, stents are substituted for saphenous vein grafts (SVG) for non-LAD lesions, and the surgical LIMA to LAD bypass is performed, ideally through a limited access, minimally traumatic approach.

Unfortunately, the published data to date on HCR must be considered limited and hypothesis generating. Clinicians, payers, and patients are interested in the specific benefits of revascularization alternatives. HCR as a scientifically validated approach would have a major healthcare impact. The ability to deliver a new therapy for CAD that provides durability, but without the obligatory trauma and prolonged recovery time characteristic of conventional CABG would be a major advance in the field of cardiovascular medicine. The NHLBI-funded Hybrid Observational Study demonstrated that equipoise exists between the two coronary revascularization paradigms; however, a rigorously designed randomized clinical trial is now needed to provide sufficient evidence to guide clinical decision making for this important patient population.

This trial is a prospective, multi-center randomized comparative effectiveness trial of HCR compared to multi-vessel PCI in patients with multi-vessel CAD involving the LAD or left main (LM) territories. The trial is designed as a "large, simple" trial, and some baseline, procedure-related and short-term outcomes data collection will be extracted from existing registry data (Society of Thoracic Surgeons [STS] Data Registry). The overall objective of this trial is to evaluate the effectiveness and safety of Hybrid Coronary Revascularization (HCR) compared to multi-vessel PCI with drug-eluting stents (DES) in patients with multi-vessel coronary artery disease involving the Left Main and/or Left Anterior Descending arteries.

The primary objective the trial is to determine whether hybrid coronary revascularization is associated with a reduction in Major Adverse Cardiac and Cerebrovascular Events (MACCE) compared to PCI with DES.

The secondary objectives are to determine the impact of HCR compared to PCI on health status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, inclusive of release of medical information, and Health Insurance Portability and Accountability Act (HIPAA) documentation (US sites)
* Age ≥ 18 years
* Clinical indication for coronary revascularization
* Coronary anatomy requiring revascularization as follows(2)

  * Multivessel CAD involving the LAD (proximal or mid) and/or LM (ostial, mid-shaft or distal) with at least 1 other epicardial coronary artery requiring treatment (LCX or RCA), OR
  * Single vessel disease involving the LAD and a major diagonal, with both requiring independent revascularization with at least one stent if randomized to HCR and stents for both the LAD and diagonal if randomized to multivessel PCI Note: If the patient qualifies based only on a LM lesion, then there must be involvement of the distal bifurcation (Medina 1,1,1) intended for treatment with a 2-stent approach (separate stents into the LAD and LCX) if randomized to PCI. However, if the patient also has non-LM disease in the RCA and/or non-ostial LAD and/or non-ostial LCX that requires separate treatment, any LM lesion is a valid criterion for enrollment, whether LM ostial, shaft or distal bifurcation disease, and any strategy of treating the LM may be employed, including not treating the ostial LCX, a provisional approach or a planned 2-stent strategy as appropriate. Similarly, if the patient qualifies based only on LAD-Dg disease, whether a bifurcation lesion or separate lesions in the LAD and Dg, without RCA or LCX disease, then both the LAD and Dg must be true lesions intended for stents (planned 2-stent approach). However, if the patient has LAD-Dg disease and a lesion in the RCA or LCX that also requires treatment, the LAD-Dg disease can then be treated in any fashion (2-stents, a provisional approach, or the Dg not even dilated if it is small), according to operator preference
* Suitable candidate for both PCI with metallic DES and HCR as determined by clinical assessment and angiogram review by an interventional cardiologist and a cardiac surgeon at the enrolling clinical site
* Ability to tolerate and no plans to interrupt dual anti-platelet therapy for ≥ 6 months if presentation with stable CAD, or ≥ 12 months if presentation with biomarker positive acute coronary syndrome (ACS)
* Willing to comply with all protocol required follow-up

Exclusion Criteria:

* Previous cardiac surgery of any kind, including CABG
* Previous thoracic surgery involving the left pleural space
* Previous LM or LAD stent (a) with evidence of in-stent restenosis or (b) within 1 cm of a qualifying lesion
* Previous PCI of the LM and/or LAD within 12 months prior to randomization
* PCI with bare metal stent (BMS) within 12 months prior to randomization
* Any complication or unsuccessful revascularization with PCI within 30 days prior to randomization.

Note: A patient may be considered eligible for enrollment if PCI with DES in non-LM and non-LAD territory was performed within 30 days prior to randomization, as long as revascularization was successful and uncomplicated, or has been performed more than 30 days prior even if unsuccessful or complicated

* Planned treatment with bioresorbable vascular scaffold(s) after randomization
* Total occlusion (TIMI 0 or 1 flow) of the LM, LAD or LCX.
* Cardiogenic shock at time of screening
* STEMI within 72 hours prior to randomization
* Need for concomitant vascular or other cardiac surgery during the index hospitalization (including, but not limited to, valve surgery, aortic resection, left ventricular aneurysmectomy, and carotid endarterectomy or stenting)
* Indication for chronic oral anticoagulation therapy at the time of randomization
* Any prior lung resection
* End-Stage Renal Disease (ESRD) on dialysis
* Patients who could not be switched from prasugrel or ticagrelor to clopidogrel, should that be needed prior to a CABG, during reverse HCR
* Extra-cardiac illness that is expected to limit survival to less than 5 years
* Allergy or hypersensitivity to any of the study drugs or devices used in the trial
* Therapy with an investigational drug, device or biologic within 1 year prior to randomization, or plan to enroll patient in additional investigational study during participation in this trial
* Unable to give informed consent or potential for noncompliance with the study protocol in the judgment of the investigator
* Pregnant at time of screening or unwilling to use effective birth control measures while dual antiplatelet therapy is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Bagiella, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Alan Moskowitz, MD, Principal Investigator — Ichan School of Medicine at Mount Sinai; John Puskas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Gregg Stone, MD, Principal Investigator — Columbia University
Locations (46):
- United States (39):
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - Yale University, New Haven, Connecticut
  - HealthPark Lee Memorial Health Systems, Fort Myers, Florida
  - Orlando Health Heart Institute, Orlando, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Maryland, College Park, Maryland
  - Universty of Minnesota, Minneapolis, Minnesota
  - Our Lady of Lourdes Medical Center, Camden, New Jersey
  - Buffalo General Medical Center/Gates Vascular Institute, Buffalo, New York
  - Mount Sinai Beth Israel, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St. Joseph's Hospital Health Center, Syracuse, New York
  - Montefiore - Einstein, The Bronx, New York
  - Duke University, Durham, North Carolina
  - WakeMed Health and Hospitals, Raleigh, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Pinnacle Health Cardiovascular System, Harrisburg, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - The Reading Health System, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Research Institute at The Heart Hospital Baylor Plano, Plano, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Gundersen Health System, La Crosse, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Centre Intégré Universitaire/Sacre Coeur, Montreal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ganyukov VI, Kochergin NA, Shilov AA, Tarasov RS, Skupien J, Kozyrin KA, Barbarash OL, Musialek P. Randomized Clinical Trial of Surgical Versus Percutaneous Versus Hybrid Multivessel Coronary Revascularization: 3 Years' Follow-Up. JACC Cardiovasc Interv. 2021 May 24;14(10):1163-1165. doi: 10.1016/j.jcin.2021.02.037. No abstract available. PMID 34016423

RESULTS

PARTICIPANT FLOW:
Groups:
- Hybrid Coronary Revascularization Group: Hybrid Coronary Revascularization (HCR) is defined, for the purposes of this trial, as a planned off-pump minimally invasive (sternal-sparing), isolated LIMA-LAD revascularization, combined with percutaneous revascularization of at least one non-LAD target.
  Hybrid Coronary Revascularization (isolated LIMA-LAD): sternal-sparing, off-pump, isolated LIMA-LAD revascularization
  Hybrid Coronary Revascularization (PCI): percutaneous revascularization of at least one non-LAD target
Period: Overall Study
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Started | 88 | 112
Completed | 61 | 71
Not Completed | 27 | 41
Not completed — Death | 4 | 9
Not completed — Lost to Follow-up | 21 | 30
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention | Total
Number analyzed (Participants) | 88 | 112 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (8.8) | 66.8 (9.2) | 65.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 36 | 61
  Male | 63 | 76 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 22 | 44
  Not Hispanic or Latino | 66 | 84 | 150
  Unknown or Not Reported | 0 | 6 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 12 | 15 | 27
  White | 67 | 78 | 145
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 12 | 17
New York Heart Association (NYHA) Classification [Count of Participants; unit: Participants] — Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients. Population: NYHA denominators differ from the overall study population due to missing data.
  Participants
    No Heart Failure: number analyzed (Participants) | 86 | 110 | 196
    No Heart Failure | 38 | 41 | 79
    Class I: number analyzed (Participants) | 86 | 110 | 196
    Class I | 18 | 23 | 41
    Class II: number analyzed (Participants) | 86 | 110 | 196
    Class II | 20 | 28 | 48
    Class III: number analyzed (Participants) | 86 | 110 | 196
    Class III | 5 | 13 | 18
    Class IV: number analyzed (Participants) | 86 | 110 | 196
    Class IV | 5 | 5 | 10
Angina Class - CCSC [Count of Participants; unit: Participants] — Grade I - Ordinary physical activity does not cause angina, such as walking and climbing stairs. Angina with strenuous or rapid or prolonged exertion at work or recreation Grade II - Slight limitation of ordinary activity. Grade III - Marked limitation of ordinary physical activity. Walking one or two blocks on the level and climbing one flight of stairs in normal conditions and at normal pace Grade IV - Inability to carry on any physical activity without discomfort, anginal syndrome may be present at rest Population: CCSC denominators differ from the overall study population due to missing data.
  Participants
    No Angina: number analyzed (Participants) | 88 | 110 | 198
    No Angina | 26 | 27 | 53
    Grade I: number analyzed (Participants) | 88 | 110 | 198
    Grade I | 11 | 17 | 28
    Grade II: number analyzed (Participants) | 88 | 110 | 198
    Grade II | 19 | 22 | 41
    Grade III: number analyzed (Participants) | 88 | 110 | 198
    Grade III | 27 | 30 | 57
    Grade IV: number analyzed (Participants) | 88 | 110 | 198
    Grade IV | 5 | 16 | 21
SF-12 Score [Mean (Full Range); unit: units on a scale] — Short Form Survey (SF-12) is a 12-item scale. Each composite score from 0-100, with total score from 0 (lower health status) to 100 (higher health status). Population: SF-12 denominators differ from the overall study population due to missing data.
  units on a scale
    Physical Health Composite Score: number analyzed (Participants) | 86 | 111 | 197
    Physical Health Composite Score | 41.5 [16.0 to 61.0] | 42.4 [9.4 to 62.4] | 41.7 [9.4 to 62.4]
    Mental Health Composite Score: number analyzed (Participants) | 86 | 111 | 197
    Mental Health Composite Score | 53.6 [16.0 to 66.8] | 54.0 [21.4 to 69.7] | 53.9 [16.0 to 69.7]
Euroqol Health Rating [Mean (Full Range); unit: units on a scale] — The Euroqol Health Rating scores range from 0 - 100, higher score indicates better health outcome. Population: Euroqol denominators differ from the overall study population due to missing data.
  units on a scale
    number analyzed (Participants) | 86 | 112 | 198
    (all) | 75.0 [0.0 to 100.0] | 75.0 [0.0 to 100.0] | 75.0 [0.0 to 100.0]
Risk Factors [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Risk factor denominators differ from the overall study population due to missing data.
  Participants
    Diabetes: number analyzed (Participants) | 87 | 111 | 198
    Diabetes | 50 | 54 | 104
    Dyslipidemia: number analyzed (Participants) | 87 | 111 | 198
    Dyslipidemia | 77 | 88 | 165
    Hypertension: number analyzed (Participants) | 87 | 111 | 198
    Hypertension | 72 | 99 | 171
    Dialysis: number analyzed (Participants) | 87 | 111 | 198
    Dialysis | 1 | 2 | 3
    Tobacco Use: number analyzed (Participants) | 87 | 108 | 195
    Tobacco Use | 19 | 10 | 29
    Lung Disease: number analyzed (Participants) | 85 | 107 | 192
    Lung Disease | 13 | 12 | 25
    Liver Disease: number analyzed (Participants) | 87 | 111 | 198
    Liver Disease | 5 | 2 | 7
    Immunocompromise Present: number analyzed (Participants) | 87 | 111 | 198
    Immunocompromise Present | 5 | 3 | 8
    Peripheral Artery Disease: number analyzed (Participants) | 87 | 111 | 198
    Peripheral Artery Disease | 4 | 5 | 9
    Cerebrovascular Disease: number analyzed (Participants) | 85 | 109 | 194
    Cerebrovascular Disease | 11 | 5 | 16
    Previous PCI: number analyzed (Participants) | 87 | 111 | 198
    Previous PCI | 37 | 44 | 81
    Previous MI: number analyzed (Participants) | 81 | 108 | 189
    Previous MI | 34 | 42 | 76
    Heart Failure: number analyzed (Participants) | 83 | 109 | 192
    Heart Failure | 10 | 25 | 35
    Arrhythmia: number analyzed (Participants) | 83 | 110 | 193
    Arrhythmia | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Coronary and Cerebrovascular Events (MACCE)
Description: The current sample size of 200 patients will not provide sufficient power to test the original null hypothesis of the trial. However, it will allow for an estimate of the MACCE rate in the two groups. A 2-year follow-up will be used to capture and understand the difference in MACCE between the two procedures. This reasoning is based on the NHLBI-funded Hybrid Revascularization Observational Study (ClinicalTrials.gov Identifier NCT01121263), which enrolled 200 HCR and 98 multi-vessel PCI with drug-eluting stent (DES) patients, and demonstrated similar risk-adjusted MACCE rates over the first 12 months following the intervention but divergence by approximately 18 months of followup.
  Therefore, it is important to continue the follow-up of the 200 randomized patients to at least 24 months. Of note, some patients who were enrolled early in the trial will have up to 3 years of follow-up data collected by the time the final patient randomized completes the 2-year time point.
Time Frame: Up to 24 months
Measure: Number (95% Confidence Interval); unit: MACCE Event Rate per Person-Year
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 88 | 112
MACCE Event Rate per Person-Year | 0.130 [0.080 to 0.211] | 0.111 [0.073 to 0.167]

2. Secondary Outcome: Hemoglobin Levels
Description: For HCR patients, lab values are pre- and post-CABG. For PCI patients, lab values are pre- and post- the last PCI.
Time Frame: Up to 90 days post-randomization
Population: The overall analysis population represents the number of patients who contributed to at least one of the pre/post measurements. Patients randomized to the HCR arm and received PCI only OR patients randomized to the PCI arm and received CABG are not included. Most patients switched interventions due to their preference. Patients who did not receive any procedures are also excluded. Patients received no interventions due to physician decision or early termination (withdrawal or lost to follow-up).
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 70 | 89
g/dL
  Pre-Procedure: number analyzed (Participants) | 66 | 87
  Pre-Procedure | 13.95 [12.80 to 15.20] | 13.40 [12.20 to 14.70]
  Post-Procedure: number analyzed (Participants) | 70 | 69
  Post-Procedure | 10.95 [9.90 to 12.30] | 12.90 [11.80 to 14.10]

3. Secondary Outcome: Creatinine Levels
Description: For HCR patients, lab values are pre- and post-CABG. For PCI patients, lab values are pre- and post- the last PCI.
Time Frame: Up to 90 days post-randomization
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 70 | 89
mg/dL
  Pre-Procedure: number analyzed (Participants) | 70 | 87
  Pre-Procedure | 0.95 [0.82 to 1.14] | 0.95 [0.81 to 1.11]
  Post-Procedure: number analyzed (Participants) | 70 | 73
  Post-Procedure | 1.03 [0.89 to 1.22] | 0.93 [0.80 to 1.17]

4. Secondary Outcome: CK-MB Levels (ng/dL)
Description: For HCR patients, lab values are pre- and post-CABG. For PCI patients, lab values are pre- and post- the last PCI.
Time Frame: Up to 90 days post-randomization
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 17 | 23
ng/dL
  Pre-Procedure: number analyzed (Participants) | 9 | 16
  Pre-Procedure | 0.90 [0.50 to 1.20] | 1.80 [1.15 to 3.15]
  Post-Procedure: number analyzed (Participants) | 15 | 16
  Post-Procedure | 2.79 [2.20 to 4.90] | 3.75 [2.60 to 8.30]

5. Secondary Outcome: CK-MB Levels (IU/L)
Description: For HCR patients, lab values are pre- and post-CABG. For PCI patients, lab values are pre- and post- the last PCI.
Time Frame: Up to 90 days post-randomization
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 7 | 4
IU/L
  Pre-Procedure: number analyzed (Participants) | 6 | 4
  Pre-Procedure | 72.00 [39.00 to 118.00] | 62.00 [33.00 to 96.50]
  Post-Procedure: number analyzed (Participants) | 4 | 4
  Post-Procedure | 311.00 [62.55 to 1045.00] | 77.00 [44.00 to 119.50]

6. Secondary Outcome: Troponin Levels
Description: For HCR patients, lab values are pre- and post-CABG. For PCI patients, lab values are pre- and post- the last PCI.
Time Frame: Up to 90 days post-randomization
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 45 | 69
ng/mL
  Pre-Procedure Troponin I: number analyzed (Participants) | 27 | 50
  Pre-Procedure Troponin I | 0.03 [0.01 to 0.18] | 0.03 [0.01 to 0.12]
  Post-Procedure Troponin I: number analyzed (Participants) | 37 | 46
  Post-Procedure Troponin I | 0.30 [0.13 to 0.97] | 0.17 [0.03 to 0.81]
  Pre-Procedure Troponin T: number analyzed (Participants) | 5 | 13
  Pre-Procedure Troponin T | 0.03 [0.02 to 0.31] | 0.01 [0.01 to 0.03]
  Post-Procedure Troponin T: number analyzed (Participants) | 7 | 12
  Post-Procedure Troponin T | 0.05 [0.01 to 0.34] | 0.01 [0.01 to 0.35]

7. Secondary Outcome: Number of Participants Requiring Medications
Description: For HCR patients, medications are prior/during/after CABG. For PCI patients, medications are prior/during/after the last PCI. Number of participants requiring medications at any time 24 Hours Prior to, During, and Within 24 Hours of the Procedure. Procedures can occur up to 90 days after randomization.
Time Frame: 24 Hours Prior to, During, and Within 24 Hours of the Procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 85 | 103
Participants
  Antiplatelets | 74 | 101
  Anticoagulants | 53 | 66
  Beta Blockers | 73 | 65
  ACE Inhibitors or ARBs | 22 | 37
  Diuretics | 25 | 18
  Statins | 71 | 79

8. Secondary Outcome: Number of Participants Requiring Transfusion
Description: Number of participants requiring transfusion during procedure and after procedure
Time Frame: Up to 90 days post-randomization
Population: The overall analysis population represents the number of patients who contributed to at least one of the intra/post measurements. Patients with at least one post-randomization procedure are included. Additional patients are missing data on transfusions.
Measure: Count of Participants; unit: Participants
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 69 | 109
Participants
  Transfusion Intra-Procedure | 3 | 1
  Transfusion Post-Procedure: number analyzed (Participants) | 69 | 108
  Transfusion Post-Procedure | 6 | 1

9. Secondary Outcome: Length of Stay
Description: Length of stay for all study procedures combined, beginning at date of procedure
Time Frame: Up to 90 days post-randomization
Population: Patients with at least one post-randomization procedure are included. Additional patients are missing data on length of stay.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 72 | 109
days | 7.00 [6.00 to 9.00] | 2.00 [2.00 to 4.00]

10. Secondary Outcome: Discharge Disposition
Description: Discharge disposition is for the last study procedure
Time Frame: Up to 90 days post-randomization
Population: Patients with at least one post-randomization procedure are included. Additional patients are missing data on discharge disposition.
Measure: Count of Participants; unit: Participants
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 83 | 109
Participants
  Home | 76 | 105
  Extended Care/Transitional Care Unit/Rehab | 5 | 3
  Other Acute Care Hospital | 0 | 1
  Nursing Home | 1 | 0
  Other | 1 | 0

11. Secondary Outcome: Cost-Effectiveness
Description: Health Status as measured by cost-effectiveness. Cost-effectiveness will be evaluated using a micro-simulation model, which will predict the accrued health care costs and quality-adjusted life expectancy for each subject at the end of the trial follow-up period and in addition over a lifetime horizon.
Time Frame: Up to 24 months
Population: While quality of life data was collected, they are not usable in a cost-effectiveness analysis due to the reduced sample size and reduced follow-up. In addition, since the trial was halted prematurely, cost data was not collected. Therefore, a cost-effectiveness analysis is not feasible.
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Feasibility of Incorporating Registry Data in a Randomized Clinical Trial
Description: For the HCR group, partial data will be extracted and transferred from the STS registry. Thus, this study will also allow evaluation of the process of data transfer, assessment of the data quality, and eventually determination of the feasibility to conduct a clinical trial with data linked to a registry.
Time Frame: Up to 24 months
Population: HCR: Obtaining data from the STS registry was not straightforward and was related to difficulty in obtaining the data and linking all clinical trial patients with their STS data. In general, more work needs to be done before registry data can be incorporated into clinical trials.
  PCI: Researchers were unable to obtain data from CATH-PCI registry. At the time of trial start-up, the registry was being restructured and moved to a different platform. Linkage to clinical trial data was not possible.
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Serious adverse events include components of the primary endpoint, which, according to the protocol, will be analyzed on an intent-to-treat (ITT) basis.
Arm/Group | Hybrid Coronary Revascularization Group | Percutaneous Coronary Intervention
All-Cause Mortality (participants affected / at risk) | 4/88 | 9/112
Serious Adverse Events (participants affected / at risk) | 20/88 | 11/112
Other Adverse Events (participants affected / at risk) | 18/88 | 9/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hybrid Coronary Revascularization Group (N=88) | Percutaneous Coronary Intervention (N=112)
Bleeding (Blood and lymphatic system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 3 | 3
Post-Pericardiotomy Syndrome (Cardiac disorders) | 2 | 0
Stent Thrombosis (Cardiac disorders) | 0 | 2
Graft Stenosis or Occlusion (Cardiac disorders) | 2 | 0
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 | 0
Infection Requiring Antibiotics (Infections and infestations) | 5 | 1
Ischemic Stroke (Nervous system disorders) | 1 | 0
Other Bleeding (Nervous system disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 2 | 0
Renal and Urinary Bleeding (Renal and urinary disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Unplanned Repeat Revascularization (Surgical and medical procedures) | 8 | 8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hybrid Coronary Revascularization Group (N=88) | Percutaneous Coronary Intervention (N=112)
Bleeding (Blood and lymphatic system disorders) | 0 | 2
Atrial Fibrillation (Cardiac disorders) | 6 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 2
Post-Pericardiotomy Syndrome (Cardiac disorders) | 4 | 0
Gastrointestinal Bleeding (Gastrointestinal disorders) | 3 | 1
Ischemic Stroke (Nervous system disorders) | 1 | 0
Unknown Etiology Stroke (Nervous system disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 2 | 1
Renal and Urinary Bleeding (Renal and urinary disorders) | 1 | 1
Mediastinal Bleeding (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Unplanned Repeat Revascularization (Surgical and medical procedures) | 4 | 3
Vascular Bleeding (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT03089398/Prot_SAP_000.pdf